CLINICAL TRIAL: NCT06076174
Title: Effects of 6-week Telerehabilitation Exercise Programme on Chronic Non-specific Neck Pain: a Pilot Randomized Controlled Trial
Brief Title: Effects of 6-week Telerehabilitation Exercise Programme on Chronic Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Zaina Ahmed, Graduate Teaching Assistant, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-23-02-27-01-PG
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Non-specific Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehab (Experimental): 6-week home-based exercise programme, will be monitored via the software that records each session so the therapist can review
  Interventions: Other: 6-week home-based exercise programme
- Conventional (Active Comparator): 6-week home-based exercise programme, will have written instructions on paper to follow through by participant themselves
  Interventions: Other: 6-week home-based exercise programme

INTERVENTIONS:
Other: 6-week home-based exercise programme — All participants will have an in-person session with the physiotherapist for exercise demonstration before beginning the programme. They will carry out the exercises independently at home over a period of six weeks, thrice a week, giving a total of 18 sessions, each lasting 30 minutes.

SUMMARY:
This study will be a pilot randomized controlled trial, comparing the effectiveness of two modes of delivery of the same 6-week exercise program for chronic non-specific neck pain. The first group will be monitored via the software that records each session so the therapist can review, and the second will have written instructions on paper to follow through by them themselves. Pre-test and post-test measurements (pain score, disability index, cervical ROM, cervical muscle endurance) will be taken, before and after completion of the exercise programme.

DETAILED DESCRIPTION:
Following ethical approval from UOS Research Ethics Committee, data collection will begin. E-posters will be sent out as recruitment announcement and those who willingly volunteer and fit the inclusion criteria will be selected. Once they sign the digital informed consent form, which will be created via Microsoft Forms, they will be randomized into either telerehabilitation group or conventional group.

Randomization will be done using permuted block method, with treatment allocation concealed. Baseline measurements from all participants will be obtained, by physiotherapist, prior to start of the exercise programme: VAS pain socre, NDI score, CROM (flexion, extension, lateral flexion, rotation) and cervical muscle endurance.

All participants will have an in-person session with the physiotherapist for exercise demonstration before beginning the programme. They will carry out the exercises independently at home over a period of six weeks, thrice a week, giving a total of 18 sessions, each lasting 30 minutes.

The software group will do each session via the CareSpace software that will record and store the entirety of the session on cloud giving the therapist access to review it. The conventional group will be given a flyer with written instructions. After two weeks, the physiotherapist will hold the first review session with each participant, held online face-to-face for those in the software group (via ConnectToMyDoctor application) and over the telephone for those in the conventional group. Similarly, after four weeks, the second review session will be held. Progressions for exercises will be given to the participants at both review sessions. On completion of all 6 weeks of the exercise programme, post-test measurements will be carried out.

For data analysis, The distribution of the data will be analyzed with Shapiro-Wilks's test. Descriptive analyses will be used for the calculation of frequencies, means, and standard deviations. For baseline differences between groups, independent samples t- test will be used. Repeated measures ANOVA will be used for within-group and between-group analyses at three different time points (0 week, 3 weeks, 6 weeks). A p value below 0.05 will be considered significant. Statistical analyses will done using SPSS version 26.0

ELIGIBILITY:
Inclusion Criteria:

* residents of UAE, both males and females
* aged between 18 45
* have normal BMI
* referred to physiotherapy for chronic non-specific neck pain
* minimum pain score of 3cm on the VAS
* pain onset at least 3 weeks ago
* have given informed consent for voluntary participation.

Exclusion Criteria:

* diagnosed by a physician with any pathological condition as cause of chronic neck pain
* presently undergoing any physical treatment or taking any medication for said pain
* has comorbidities, such as diabetes and hypertension
* has conditions like migraine and cervicogenic headache
* has vertigo and/or vertebrobasilar insufficiency,
* physically disabled or has recent immobilizing injury
* orthopaedic conditions, such as spondylosis, spondylolisthesis, wryneck
* history of neurological conditions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Adherence | pre and immediately post intervention, 6 weeks
  Frequency per week (Number of sessions completed each week) will be noted through exercise diary fro conventional group, and recordings on cloud for tele rehab group.
Adherence | pre and immediately post intervention, 6 weeks
  Duration of each session will be noted through exercise diary fro conventional group, and recordings on cloud for tele rehab group.

SECONDARY OUTCOMES:
Visual Analogue Scale for Pain | pre and immediately post intervention, 6 weeks
  Visual Analogue Scale for Pain (VAS Pain) is a continuous scale in the form of a 100mm line, marked by "no pain" (score of 0) on one end and "pain as bad as it could be" (score of 100) on the other end.
Neck Disability Index questionnaire | pre and immediately post intervention, 6 weeks
  It consists of 10 items, each scored from 0 - 5, giving a total out of 50, where a higher score is indicative of increased disability.
CROM instrument | pre and immediately post intervention, 6 weeks
  Cervical range of motion
Cranio-cervical Flexion Test | pre and immediately post intervention, 6 weeks
  Cervical muscle endurance assessed by therapist

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed ZZ, Khan MN, Bairapareddy KC. Randomised controlled trial assessing the effects of 6-week telerehabilitation exercise programme on chronic non-specific neck pain: a study protocol. BMJ Open Sport Exerc Med. 2024 Feb 26;10(1):e001874. doi: 10.1136/bmjsem-2023-001874. eCollection 2024. PMID 38420117